

COVER PAGE WITH THE OFFICIAL TITLE OF THE STUDY: SUITABILITY, CLINICAL UTILITY AND ACCEPTABILITY OF A TRANSDIAGNOSTIC INTERVENTION VIA THE INTERNET FOR THE TREATMENT OF EMOTIONAL DISORDERS AND THOSE DERIVED FROM STRESS AND TRAUMA.

DATE: OCTOBER 1, 2021



## INFORMED CONSENT

Dear participant, you have been invited to a scientific study with the support of PAPIIT grant IT300721, entitled: "Suitability, clinical utility and acceptability of a transdiagnostic intervention via the Internet for the treatment of emotional disorders and those derived from stress and trauma" that is carried out carried out by members of the Laboratory of Psychology and Technological Innovation (LABPSIIT) of the *Iztacala* School of Higher Studies of the National Autonomous University of Mexico. The project has the endorsement of the Ethics Commission of the *Iztacala* School of Higher Studies, UNAM (CE / FESI / 082020/1363). The purpose of this notice is to inform you of the objectives of the project as well as the confidential use of your data derived from the study.

The objective of the study is to determine the suitability, clinical utility and acceptability of an intervention program based on the transdiagnosis approach via the internet. aimed at adults who meet diagnostic criteria for an emotional disorder or derived from a stressful or traumatic event. The clinical evaluation of the users will be carried out in 4 moments (before, after and at three and six months after the treatment). The initial evaluation will be carried out by videoconference, it will consist of the application of a series of questionnaires that will help to assess your emotional distress. Once the evaluation is completed, you will be assigned to one of the study conditions (transdiagnostic treatment, cognitive behavioral therapy or waiting list). Participants in the waiting list control group will receive the intervention 2 months after the evaluation and will be assigned to the intervention that has shown the best results and satisfaction. The intervention will be carried out through the internet and will consist of between 8 and 10 sessions, a weekly session of one hour in individual online format. All participants may withdraw from treatment at any time.

The requested Personal Data will be processed for research, teaching and statistical purposes. They will be protected through a code (folio) that guarantees their confidentiality; Access to the data will be limited to the main researcher of the study and the management technician of the institutional server housed in the facilities of the Distance Education Coordination of the *Iztacala* School of Higher Studies, UNAM, with address at Av de los Reyes 1, Tlalnepantla de Baz, México CP 5700. Likewise, the data will be kept during your participation in the intervention and, once concluded, will be kept for an additional period of up to 5 years to later be eliminated in order to avoid improper treatment. thereof. By virtue of the foregoing, the information provided will be treated with all appropriate security measures, in accordance with the principles contained in the Federal Law on Protection of Personal Data Held by Private Parties, its Regulations and the Guidelines of the Privacy Notice of the United Mexican States.



## Consequences:

The risks of your participation are minimal, some questions in the questionnaires assess your mood and you could relive stressful situations, which could cause you some discomfort or emotional distress, but we ask that you answer them because they are important to the study. Likewise, during the treatment sessions you could present a greater manifestation of emotions or feelings, do not be alarmed, it is normal because the central mechanism of the intervention is emotional regulation in the face of various vicissitudes of life. If you develop acute discomfort, report it immediately to your counselor.

## Profits:

If you agree to participate, you will join a free psychological support program by supervised and qualified psychological advisors, who could be students in training from the last semesters of the Psychology career. The duration of the intervention program may vary among users depending on their treatment condition and the time available for the intervention; however, it will be arranged between 8 and 10 sessions, a weekly session of one hour in individual online format.

For more questions, you can contact us by email: labpsiit@iztacala.unam.mx

To begin, we ask you to answer a series of questionnaires that will be presented below, which will take about 25 minutes. There are no right or wrong questions, so please answer as honestly as possible.

"I have read this informed consent document; I have understood the explanations provided in it about the objective of the research project. I also understand that, at any time and without giving any explanation, I can revoke the consent that I now submit. I have also been informed and understand that the data I provide will be protected and used solely for academic and research purposes. I voluntarily consent to my participation in the intervention program under the characteristics that operate in it and that were previously mentioned. I understand that I have the right to withdraw my participation at my own will ".

You may receive a copy of this informed consent to your provided email and may request its cancellation through the following email: labpsiit@iztacala.unam.mx